CLINICAL TRIAL: NCT04956159
Title: Evaluating the Antidepressant Efficacy of Transcranial Magnetic Stimulation (TMS) in Patients With Inflammatory Bowel Disease (IBD) and Effects on IBD-related Symptoms.
Brief Title: TMS in Inflammatory Bowel Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: University of Calgary (Other)
Collaborators: IMAGINE (Inflammation, Microbiome, and Alimentation: Gastro-Intestinal and Neuropsychiatric Effects) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB20-1272
Record Dates: First submitted 2021-01-13; First posted 2021-07-09 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2021-11

CONDITIONS: Inflammatory Bowel Diseases; Maladaptive Behavior Associated With Physical Illness
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active iTBS rTMS (Active Comparator): The active arm involves magnetic stimulation of the brain to the left dorsolateral prefrontal cortex (DLPFC) twice daily for two weeks (20 sessions). The active arm will be receiving intermittent Theta-Burst (iTBS) repetitive Transcranial Magnetic Stimulation (rTMS) to deliver magnetic pulses.
  Interventions: Device: iTBS repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham iTBS rTMS (Sham Comparator): sham rTMS treatment involves scalp stimulation with no magnetic pulse twice daily for two weeks (20 sessions). Sham rTMS involves only the click replicating the sound of the magnetic discharge, without any magnetic pulse being delivered to the brain.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: iTBS repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a non-invasive procedure in which cerebral electrical activity is influenced by a rapidly changing magnetic field. The magnetic field is created by a plastic-encased coil which is placed over the patient's scalp. The magnetic field can be directed onto specific areas of the brain. rTMS can modulate cerebral activity by low or high frequencies. Over time, the magnetic field pulses can gradually change the activity level of the stimulated brain region and help symptoms of depression and anxiety.
  Other Names: MAGPRO X100 stimulator
  Arms: Active iTBS rTMS
Device: Sham rTMS — Sham rTMS involves a click replicating the sound of the magnetic discharge, without any magnetic pulse being delivered.
  Other Names: MAGPRO X100 stimulator
  Arms: Sham iTBS rTMS

SUMMARY:
Transcranial magnetic stimulation (rTMS) has demonstrated diagnostic and therapeutic potential for a number of conditions and is an approved treatment for depression. Inflammatory Bowel Disease (IBD) has a significant impact on mental health, and comorbid maladaptive behaviors and pain are highly prevalent in patients with IBD and are often under-treated.

The investigators predict TMS will improve comorbid maladaptive behavior (heightened interoceptive awareness, sleep, fatigue, catastrophizing, anxiety and depression), reduce pain and improve quality of life in persons with inflammatory bowel disease (IBD). Further, TMS benefits will be associated with changes in gut microbiome as measured by stool, blood and urine samples and normalization of IBD-associated changes in brain structure and/or function as measured by magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Background and rationale:

Comorbid maladaptive behaviors and pain are highly prevalent in patients with IBD and are often under-treated. These comorbidities lack effective therapies and thus complicate medical management, adversely impact patient outcome and health, and increase the resource burden on the healthcare system. Development of effective treatment delivery is therefore vital. Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive form of brain stimulation in which an electric pulse generator placed at the scalp produces a rapidly changing magnetic field at biologically relevant frequencies to induce a stimulating electrical current at targeted sites in the brain. rTMS has demonstrated diagnostic and therapeutic potential for a number of conditions, including Alzheimer's disease, autism, bipolar disorder, epilepsy, chronic pain, major depressive disorder, Parkinson's disease, post-traumatic stress disorder (PTSD), schizophrenia (negative symptoms), obsessive-compulsive disorder (OCD), and for the cessation of smoking. To date, however, rTMS has not been used to treat the mental health issues and symptoms observed in persons with IBD. The investigators will develop rTMS interventions for IBD to target comorbid maladaptive behaviors and pain using evidence-based knowledge of TMS effectiveness for other chronic medical conditions.

Research Question:

Compared to sham, does twice daily intermittent theta-burst stimulation rTMS delivered to the left dorsolateral prefrontal cortex for two weeks (20 sessions) improve comorbid maladaptive behavior (heightened interoceptive awareness, sleep, fatigue, catastrophizing, anxiety and depression), reduce pain and improve quality of life in persons with inflammatory bowel disease (IBD)? Further, will TMS benefits be associated with changes in gut microbiome and normalization of IBD-associated changes in brain structure and/or function as measured by magnetic resonance imaging (MRI)?

Methods:

Forty male and female IBD (Chron's Disease (CD) and Ulcerative Colitis (UC)) patients with co-morbid anxiety and depression will be recruited for this study.

Patients will be randomized 1:1 to TMS or sham TMS according to a computer-generated randomization list from eligible patients identified from the cohort study. Randomization will be stratified by type of IBD (UC versus CD). Patients will be randomized 1:1 to 2 weeks of twice-daily active or sham TMS. The investigators will utilize intermittent theta-burst stimulation (iTBS 600 pulses per session delivered as triplets at 50Hz repeated at 5Hz at 80% resting motor threshold) delivered to the left dorsolateral prefrontal cortex (DLPFC) using a MagPro X100 stimulator and a COOL-B70 (active) or MCF-P-B70 (placebo) coil. Participants will receive 20 treatments over two weeks. All participants allocated to the double-blind phase will be offered 2 weeks of open-label twice-daily iTBS to the left DLPFC if they do not achieve 50% reduction in QIDS-SR score during the double-blind phase.

Baseline characterization will include demographic information, self-reported measures of comorbid maladaptive behaviors and pain, neurocognitive tests, analysis of IBD symptoms, microbiome analysis

Participants will undergo an MRI of the brain prior to receiving treatment for localization of the DLPFC, as well as characterization of volumetric imaging, white matter imaging, resting state activity and inflammation imaging. A second MRI will be repeated characterizing these same parameters after the conclusion of the sham-controlled treatment (week 2).

Stool, blood and urine samples will be collected at baseline, after the conclusion of the sham-controlled treatment (week 2) and 4 weeks follow up (week 6). These will be used for assessment of fecal calprotectin, fecal bacterial and fungal microbiome, inflammatory markers and metabolomic analysis.

Brief, computerized neurocognitive tests will be administered at baseline, after TMS treatment (week 2) and 4 week follow up (week 6)

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of IBD, demonstrated to be in endoscopic remission (Mayo Endoscopic Subscore [for UC] 0 or 1, or Simple Endoscopic Score for CD ≤4) or biomarker remission (fecal calprotectin <250 ug/g) within 6 months of randomization
* ≥8 on the Hospital Anxiety and Depression Scale
* on stable IBD-related and psychotropic medications for the four weeks preceding randomization

Exclusion Criteria:

* severely active IBD (Mayo score > 9, HBI > 16)
* require systemic corticosteroids
* initiated biologic treatment within the preceding three months
* suicidal ideation
* psychosis
* having failed ECT
* previous rTMS treatment (for blinding integrity)
* contraindications for MRI
* Use of benzodiazepines or GABA agonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Change in depressive and anxiety symptoms with active iTBS-rTMS as compared to sham treatment group | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  Hospital Anxiety and Depression Scale (HADS) will be used to assess anxiety and depression. The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.

SECONDARY OUTCOMES:
Change in depressive symptoms as measured by Montgomery-Åsberg Depression Rating Scale (MADRS) score from baseline to week-2 (post rTMS treatment) with iTBS-rTMS as compared to sham treatment group | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. Compared to sham-rTMS, active-iTBS rTMS is anticipated to show Higher rates of clinical remission (score ≤12 on the MADRS) and Higher rates of clinical response (≥50% reduction in MADRS scores)
Change in mood from baseline to week 2 (post rTMS treatment) with iTBS-rTMS as compared to sham treatment group | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  Young Mania Rating Scale (YMRS) will be used to assess changes in mood from baseline to Week 4. The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in manic symptoms. Total score ≤12 indicates remission (13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania)
Change in IBD symptoms with active iTBS rTMS compared to sham rTMS | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  The Short Inflammatory Bowel Disease Questionnaire (short IBDQ) will be used to measure symptoms of persons with inflammatory bowel disease. The minimum score for Short IBDQ is 10 points, indicating very poor quality of life, while the maximum score is 70 points, indicating an optimal quality of life.
Change in quality of life in persons with IBD with active iTBS rTMS compared to sham rTMS | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  The EuroQol-5 Dimension-5 Level (EQ-5D-5L) is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).
Change in self reported anxiety symptoms in persons with IBD with active iTBS rTMS compared to sham rTMS | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  The General Anxiety Disorder 7-item scale (GAD-7) is a tool for self reported measure of patient anxiety. Scores range from 0 (no anxiety) to 35 (severe anxiety) with scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Change in self reported depressive symptoms in persons with IBD with active iTBS rTMS compared to sham rTMS as measured by the Patient Health Questionaire. | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  The Patient Health Questionaire-9 (PHQ-9) is a 9-item questionnaire which objectifies degree of depression severity. Scores range from 0-4 = no depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19= moderately severe depression, 20-27 = severe depression.
Change in self reported depressive symptoms in persons with IBD with active iTBS rTMS compared to sham rTMS as measured by the Quick Inventory of Depressive Symptomatology | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  The Quick Inventory of Depressive Symptomatology (QIDS) rates depression symptoms via self-assessment.Severity of depression can be judged based on the total score.
  1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression
Change in self reported physical, mental and social health and well-being in persons with IBD with active iTBS rTMS compared to sham rTMS | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  The Patient-Reported Outcomes Measurement Information System (PROMIS) is a flexible set of tools designed to measure self-reported physical, mental and social health and wellbeing. The PROMIS-29, a generic health-related quality of life survey, assesses 7 domains (depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; and ability to participate in social roles and activities) with 4 questions. The questions are ranked on a 5-point Likert Scale. There is also one 11-point rating scale for pain intensity
Change in self reported symptoms of gastrointestinal pain in persons with IBD with active iTBS rTMS compared to sham rTMS | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  The Patient-Reported Outcomes Measurement Information System (PROMIS) is a flexible set of tools designed to measure self-reported physical, mental and social health and wellbeing. The PROMIS-V10 is a brief questionnaire that asks patients 5 questions regarding belly pain during the past week. Each question is ranked on a 5-point Likert Scale, with 1 representing no symptoms and 5 representing maximal symptoms. Summation of the points gives a total score.
Change in interoceptive awareness with active iTBS rTMS compared to sham rTMS in persons with IBD. | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item state-trait questionnaire to measure multiple dimensions of interoception by self-report. Individuals rate items based on a 6 point Likert scale from 0-5 with '0' indicating 'Never' and '5' indicating 'Always'. Higher total scores and subscale scores indicate higher levels of positive awareness.
Change in catastrophizing thoughts and feelings in persons with IBD with active iTBS rTMS compared to sham rTMS | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  The Pain Catastrophizing scale is one of the most widely used instruments for measuring catastrophic thinking related to pain. People are asked to indicate the degree to which they have thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness.
Change in quality of sleep with active iTBS rTMS compared to sham rTMS in persons with IBD. | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions to measure sleep quality. The 19 self-rated items are combined to form component scores, each of with has a range of 0 (no difficulty) to 3 (severe difficulty) points. A global score of all components range from 0 (no difficulty in all areas) - 21 (severe difficulty in all areas)
Change in self reported fatigue in persons with IBD with active iTBS rTMS compared to sham rTMS | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  The Fatigue Severity Scale (FSS) is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle.
Change in cognitive function with active iTBS rTMS compared to sham rTMS in persons with IBD. | tests will also be administered at baseline and at the conclusion of the 2 week double-blind phase, and at 4 weeks post treatment (week 6)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes 4 objective cognitive tests (adapted from choice reaction time, 1-back working memory task, symbol digit coding, and Trails-B) and a subjective cognitive questionnaire (PDQ-5). Results indicate cognitive performance compared to healthy age-, sex- and education-matched individuals.
Stool samples- Individual microbial analysis | Stool will be collected at baseline, at the conclusion of the 2 week double-blind phase, and at 4 weeks post treatment (week 6)
  The investigators will assess fecal microbial diversity and the relative abundance of bacterial and fungal taxa using phyloseq along with additional R-based computational tools. Principal Component Analysis (PCoAs) will be conducted on both a variance stabilization transformed and rarefied OTU matrices and then statistically confirmed by a PERMANOVA. The Shannon and Chao1 alpha-diversity indices will be calculated using phyloseq and statistically confirmed by Mann-Whitney (GraphPad Prism software, version 5c). The R packages DESeq2 and MaAsLin will used to calculate differentially abundant microbial taxa. Correlation analysis between taxa and metadata will performed using the by bicor method in R package 'microbiome'.
Stool samples- Microbial community measurements | Stool will be collected at baseline, at the conclusion of the 2 week double-blind phase, and at 4 weeks post treatment (week 6)
  In addition to the specific microbiome analysis, composite measures using supervised (partial least squares discriminant analysis- PLS-DA) and unsupervised PCoA data reduction techniques will be explored in order to determine the most discriminatory combination of microbiome parameters. Receiver operator characteristics and permutation testing will be used to quantify discrimination performance and statistical significance, and leave-one-out-cross-validation will be used to estimate discrimination performance.
16S and ITS2 rRNA gene sequencing. | Stool, urine, and blood samples will be collected at baseline, at the conclusion of the 2 week double-blind phase, and at 4 weeks post treatment (week 6)
  The investigators aim to attempt to identify microbial biodiversity measures that best predict general anxiety, depression and pain scores and neuroimaging findings.
  All samples will be amplified by polymerase chain reaction (PCR) in triplicate using 37-nucleotide barcoded primer pairs flanking the V4 region of the 16S gene and the ITS2 gene. Pooled PCR amplicons will be sequenced across the hyper-variable regions. Sequences will be pre-processed, denoised, and quality filtered by size using DADA229. Representative sequences will be clustered into operational taxonomic units (OTUs) and classified against the Greengenes Database30 according to 97% similarity.
  Using the sequencing data, the investigators will identify the microbial features (taxa and diversity measurements) that associate with general anxiety and depression and pain scores and neuroimaging findings using methods from community ecology.
Implicit Suicidal Thoughts | tests will also be administered at baseline, at the conclusion of the 2 week double-blind phase, and at 4 weeks post treatment (week 6)
  Death Implicit Association Test (D-IAT) is a behavioral test that measures the strength of automatic (implicit) associations between concepts in people's minds relying on latency measures in a simple sorting task. The strength of an association between concepts of "death" and "ones self" is measured by the standardized mean difference score of the 'hypothesis-inconsistent' pairings and 'hypothesis-consistent' pairings
Functional Magnetic Resonance Imaging (fMRI) | Subjects will undergo MRI at 0 (baseline) and at the completion of the blinded phase (week 2)
  Change in task and resting state functional connectivity as determined by an fMRI. A whole-brain resting-state fMRI scan to determine the strength of functional connections between brain regions (inferred from degree of temporal synchrony, called connectivity) as well as the magnitude of spontaneous neuronal activity within brain regions (T2*-weighted gradient-echo echo planar imaging, 3 mm3 resolution, 2-sec temporal resolution; 8min).
Magnetic Resonance (MR) spectroscopy | Subjects will undergo MRI at 0 (baseline) and at the completion of the blinded phase (week 2)
  Change in brain metabolites in regions of interest.
Magnetic Resonance Imaging (MRI)- Volumetric imaging. | Subjects will undergo MRI at 0 (baseline) and at the completion of the blinded phase (week 2)
  Change in volume measurements in brain regions of interest. A whole-brain anatomical scan at 1 mm3 resolution to permit precise volume measurements of brain regions (3D T1-weighted; 5 min)
Magnetic Resonance Imaging (MRI)- White matter imaging | Subjects will undergo MRI at 0 (baseline) and at the completion of the blinded phase (week 2)
  Change in structural integrity of white matter tracts. A whole-brain diffusion tensor imaging (DTI ) scan to permit quantitative measurements of structural integrity within known white matter tracts (30 gradient directions, b1 = 1000, b2 = 2000 s/mm2, 2 mm3 resolution; 9 min).
Magnetic Resonance Imaging (MRI)- Inflammation imaging. | Subjects will undergo MRI at 0 (baseline) and at the completion of the blinded phase (week 2)
  Change in inflammation in brain regions of interest. A whole-brain quantitative susceptibility mapping (QSM) scan to infer the degree of inflammation within brain regions (T2*-weighted gradient-echo susceptibility weighted imaging, 8 echoes, 1 mm3 resolution; 5 min)

OTHER OUTCOMES:
Side Effects | Measured at baseline, halfway through rTMS treatment (week 1), end of rTMS treatment (week 2) and 4 weeks post treatment (week 6)
  Side effects will be tracked through the Toronto Side Effects Scale (TSES). The TSES is a self reported questionnaire that assesses incidence, frequency, and severity of central nervous system, gastrointestinal, and sexual side effects within the past 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada